CLINICAL TRIAL: NCT01847534
Title: Supplemental Parenteral Nutrition in Critically Ill Adults: A Pilot Randomised Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ANZIC RC AD 003
Record Dates: First submitted 2013-04-22; First posted 2013-05-07 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Organ Failure; Critical Illness
MeSH Terms: conditions — Multiple Organ Failure; Critical Illness | interventions — Dietary Supplements; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): Standard care: Nutrition will be managed as per best practice and local policy including the use of small bowel feeding tubes, prokinetics and PN if required to meet nutrition needs.
  Interventions: Other: Standard Care
- Supplemental PN (Experimental): Supplemental PN to complete inadequate EN provision
  1. Patients allocated to the supplemental PN (intervention) group will have PN commenced within 2 hours of randomisation. The starting dose of PN will be determined by the amount of energy received in the 24 hours prior to randomisation.
  2. EN will be managed as per local protocol however EN must not be reduced based on the supplemental PN being administered.
  3. The adequacy of nutrition provision from both PN and EN will be assessed at midday each day for 7 days or until ICU discharge. The dose of PN will be adjusted according to a prespecified schedule.
  Interventions: Other: Supplemental PN

INTERVENTIONS:
Other: Supplemental PN
  Arms: Supplemental PN
Other: Standard Care
  Arms: Standard Care

SUMMARY:
One of the essential treatments for assisting patients in their recovery from illness is the provision of nutrition in a liquid form which is delivered into the stomach or as a fluid into the vein. Until recently the benefits of nutrition were undervalued in the critically ill, however, it has now become clear that targeted nutrition can positively affect a person's outcome. This is particularly important for patients who are significantly unwell and require increased amounts of nutrition to support recovery. Inadequate nutrition therapy leads them to rapidly lose weight, predominantly in the form of muscle loss which greatly contributes to their poor recovery.

Whilst nutrition is essential for recovery, there are several issues with the delivery of nutrition via the stomach (the most commonly used method of delivering nutrition in the critically ill). For many reasons, patients are unable to tolerate large quantities of nutrition via the stomach and in addition to this there are hospital or procedural reasons for nutrition being turned off for lengthy periods of time. As such, this results in patients being delivered only about half of the nutrition that is planned. One potential way to overcome this is to deliver nutrition via the vein, whilst nutrition into the stomach continues, with the aim to meet the energy gap that is lost by inadequate nutrition via the stomach.

In this study of 100 patients, we will deliver combined nutrition via the vein and stomach in 50 patients and the other 50 patients will receive nutrition as per normal practice. We will measure important outcomes for these patients to determine if this allows us to meet significantly more of their nutrition needs. This study will also help us determine how best to design a larger study of this strategy.

DETAILED DESCRIPTION:
The principal objectives are:

1. To determine whether the supplemental Parenteral Nutrition (PN) strategy leads to the delivery of increased amounts of total nutrition (measured as energy delivered), and is safe in regards to adverse effects.
2. To measure the clinical outcomes in patients receiving both study strategies to provide information to assist design of a larger randomized controlled trial.

   Secondary objectives in a sub-set of patients are:
3. To determine whether the supplemental PN strategy leads to improved nitrogen balance.
4. To determine both the nutritional requirements and nutritional intake of critically ill patients during the period of hospitalization after transfer from the Intensive Care Unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

Patients in intensive care who meet all of the following:

* Admitted to intensive care between 48 hours and 72 hours previously
* Mechanically ventilated at the time of enrollment and expected to remain ventilated until the day after tomorrow
* At least 16 years of age
* Have central venous access suitable for PN solution administration
* Have 1 or more organ system failure (respiratory, cardiovascular or renal) related to their acute illness defined as:

  1. Partial pressure of oxygen (PaO2) / Fraction of Inspired oxygen (FiO2) ratio ≤ 300 mmHg
  2. Currently on 1 or more continuous vasopressor infusion which were started at least 4 hours ago at a minimum dose of :

     1. Dopamine greater than 5 mcg/kg/min
     2. Noradrenaline ≥ 0.1mcg/kg/min
     3. Adrenaline ≥ 0.1 mcg/kg/min
     4. Any dose of total vasopressin
     5. Milrinone >0.25mcg/kg/min)
  3. Renal dysfunction defined as

     In patients without known renal disease:
     1. serum creatinine > 171 mmol/l OR
     2. Currently receiving renal replacement therapy

        In patients with known renal disease:
     3. an absolute increase of > 50% in creatinine from baseline OR
     4. Currently receiving renal replacement therapy
  4. Currently has an intracranial pressure monitor or ventricular drain in situ
  5. Currently receiving extracorporeal membrane oxygenation
  6. Currently has a ventricular assist device

Exclusion Criteria:

* Both EN and PN cannot be delivered at enrollment (i.e. either an enteral tube or a central venous catheter cannot be placed or clinicians feel that EN or PN cannot be safely administered due to any other reason).
* Currently receiving PN
* Standard PN solutions cannot be delivered at enrolment (i.e. clinicians believe that a patient definitely needs a specific parenteral nutrition formulation (e.g. glutamine-supplementation or specific lipid formulation).
* Death is imminent or deemed highly likely in the next 96 hours.
* There is a current treatment limitation in place or the patient is unlikely to survive to 6 months due to underlying illness
* More than 80% of energy requirements have been satisfactorily delivered via the enteral route in the last 24 hours.
* Are known to be pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Total energy amount delivered | First 7 days of the study period
  The primary outcome for this pilot study is the total energy amount delivered from nutrition therapy (ie. from Enteral Nutrition (EN) and from supplemental PN, if delivered) over the first 7 days of the study period.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (2):
  - The Alfred Hospital, Melbourne, Victoria
  - Geelong Hospital, Geelong
- New Zealand (4):
  - Auckland City Hospital (CVICU), Auckland
  - Auckland City Hospital (DCCM), Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington

REFERENCES:
- [Derived] Ridley EJ, Davies AR, Parke R, Bailey M, McArthur C, Gillanders L, Cooper DJ, McGuinness S; Supplemental Parenteral Nutrition Clinical Investigators. Supplemental parenteral nutrition versus usual care in critically ill adults: a pilot randomized controlled study. Crit Care. 2018 Jan 23;22(1):12. doi: 10.1186/s13054-018-1939-7. PMID 29361959
- [Derived] Ridley EJ, Davies AR, Parke R, Bailey M, McArthur C, Gillanders L, Cooper DJ, McGuinness S; Supplemental Parenteral Nutrition Clinical Investigators. Supplemental parenteral nutrition in critically ill patients: a study protocol for a phase II randomised controlled trial. Trials. 2015 Dec 24;16:587. doi: 10.1186/s13063-015-1118-y. PMID 26703919